CLINICAL TRIAL: NCT01687738
Title: Lung Cancer Surgery: Decisions Against Life Saving Care - The Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: East Carolina University (Other); University of South Carolina (Other)
Responsible Party: Principal Investigator, Samuel Cykert, MD, Professor of Medicine and Associate Director, Medical Education, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0992; 121218-RSG-05-217-05-CPPB (Other: American Cancer Society)
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non small cell lung cancer; health disparities
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Communication Intervention (Experimental): Specially trained communicator addresses factual understanding and elicits other barriers to care
  Interventions: Other: communication intervention
- Real Time Registry and data feedback only (Experimental): Patients are enrolled in registry and clinicians receive warnings about delayed or missed care.
  Interventions: Other: Real Time Registry and data feedback only

INTERVENTIONS:
Other: communication intervention — Because of the gaps between documented outcomes of lung cancer surgery and patient communication barriers identified in our recent work, our communication intervention will focus on improving presentation of risk information and confirmation of understanding of patient medical.
  Arms: Communication Intervention
Other: Real Time Registry and data feedback only — This group of patients will not received the enhanced communication intervention
  Arms: Real Time Registry and data feedback only

SUMMARY:
Purpose: Overall lung surgery rates and black/white disparities have not improved during a decade of documentation. The goal of this study is to incorporate lessons from the previous prospective cohort study to optimize lung cancer surgery rates and narrow black-white disparities for patients diagnosed with stage I or II, non-small cell lung cancer.

Participants: Stage I and II, non-small cell lung cancer at 3 participating sites. Procedures: Phase I of the study has been completed. Phase I was a deidentified 3-year, retrospective chart review, used to establish the baseline surgical rates for the intervention. The patient enrollment phase of the study will move forward that will include use of a real time registry to follow patient progression through clinical follow up, diagnostic testing and treatment for biopsy proven or highly probable early stage, non-small cell lung cancer. The patient enrollment portion of the study will start, September 2012. All patients with Stage I or II non-small cell lung cancer who enroll in the study will be entered into real time registries at every site. Patients' progress through the registries including follow-up provider visits, diagnostic tests, and procedures will be transparent and any missed appointments will be flagged. Feedback will be given to lung cancer providers in both arms. The randomized trial will compare patients who receive usual care plus the registry to those who receive the registry plus visits and calls from a trained cancer communicator -educator (CCE) who is well versed in issues specific to lung cancer and trained in active listening and communication that accounts for patients' limitations in health literacy. The CCE will also use Kleinman's Patient Model to identify attitudes or beliefs that represent barriers to recommended care that could potentially be addressed through negotiation and more targeted communication.

The hypothesis is that an electronic warning system, data transparency, and enhanced communication will optimize lung surgery rates and reduce racial gaps.

DETAILED DESCRIPTION:
Note that the registry intervention will be compared to historical controls obtained from the electronic chart review. The main outcome will be receipt of lung resection surgery and this outcome will be assessed controlling for age, race, education, income, perceptions of communication, co-morbid illnesses, and level of health literacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or greater;
2. A probability of 60% or higher of a lung lesion being malignant as calculated by a Bayesian algorithm using clinical and radiographic characteristics or biopsy proven disease; and
3. The patient has been clinically classified as having stage I or II disease.

Exclusion Criteria:

1. incarceration / ward of the state status,
2. Severe cognitive impairment. If a patient meets the inclusion criteria but is consistently unable to comprehend survey questions during the interview process, we will exclude that patient from the overall study.
3. absolute contraindications by pulmonary function testing (FEV-1 < 25% of predicted)
4. Non-English speaking. Hispanic patients represent less than 4 percent of lung cancer patients in North Carolina restricting our ability to document an intervention effect.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2012-08; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with stage I and II, non-small cell lung cancer who receive surgery. | Baseline to 4 months
  The primary outcome variable, surgery yes or no, will be compared in the control group randomized to usual care, to the intervention group randomized to the cancer communicator.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Cykert, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Cykert S, Eng E, Walker P, Manning MA, Robertson LB, Arya R, Jones NS, Heron DE. A system-based intervention to reduce Black-White disparities in the treatment of early stage lung cancer: A pragmatic trial at five cancer centers. Cancer Med. 2019 Mar;8(3):1095-1102. doi: 10.1002/cam4.2005. Epub 2019 Feb 4. PMID 30714689

DOCUMENTS (2):
  • Study Protocol (2011-05-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT01687738/Prot_000.pdf
  • Statistical Analysis Plan (2011-05-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT01687738/SAP_001.pdf